CLINICAL TRIAL: NCT04521725
Title: Effect of Additional Monitoring Devices on Healthcare Provider Mental Workload, Visual Attention, and Performance During Neonatal Resuscitation
Brief Title: Effect of Monitoring Devices on Healthcare Provider Performance During Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Pro00097797
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Prematurity
Keywords: Neonatal resuscitation; Human Factors; Workload; Respiratory Function Monitoring; cerebral near infrared spectroscopy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1: ECG+SpO2 only (No Intervention): Traditional ECG (heart rate) and SpO2 (pulse oximetry) monitoring for resuscitation only.
- Group 2: ECG+SpO2+RFM (Active Comparator): Addition of Respiratory Function Monitor to ECG and SpO2 during resuscitation.
  Interventions: Device: Respiratory Function Monitor (RFM)
- Group 3: ECG+SpO2+RFM+NIRS (Active Comparator): Addition of cerebral NIRS and Respiratory Function Monitor to ECG and SpO2 during resuscitation.
  Interventions: Device: Respiratory Function Monitor (RFM); Device: Cerebral Near-Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Respiratory Function Monitor (RFM) — Use of respiratory function monitor to detect tidal volume and expired CO2 to guide mask ventilation during neonatal resuscitation.
  Arms: Group 2: ECG+SpO2+RFM; Group 3: ECG+SpO2+RFM+NIRS
Device: Cerebral Near-Infrared Spectroscopy (NIRS) — Use of cerebral NIRS to determine cerebral oxygenation to guide oxygen titration during neonatal resuscitation.
  Arms: Group 3: ECG+SpO2+RFM+NIRS

SUMMARY:
Babies born very early (at less than 32 weeks) usually need help to breath right at birth, also called neonatal resuscitation. Healthcare providers (HCPs) are specially trained to provide this help. HCPs uses information about the baby's condition, such heart rate and oxygen levels, to decide whether they giving the baby effective help, or whether other actions are needed. It can be very stressful for even experienced HCPs to interpret all this data, coordinate a team, make decisions, and perform specialized skills all at the same time.

More recently, new ways of monitoring how a baby is doing neonatal resuscitation has been studied. Respiratory function monitoring (RFM) is a machine that can measure how much air is going into the lungs. This is important as too much air can lead to lung damage, while too little air means that the baby isn't breathing effectively. Another measure is called cerebral near-infrared spectroscopy (cNIRS), which measures oxygen levels in the brain using a probe placed on the forehead. Providing the right amount of oxygen to the most vulnerable organ - the brain - can be important in lowering the risk for injuries to the brain such as brain bleeding. While these machines give us more information, it can also make it even harder for HCPs to focus on the task, adding more complexity to making decisions, adding to their workload, and causing more stress.

To study the effect RFM and cNIRS may have on how affects HCPs workload and stress, the investigators will study HCPs self-reported workload during three time periods - first, doing resuscitations only using basic information (Group 1: heart rate, oxygen levels, direct observations of the baby), second, adding RFM (Group 2), finally adding both RFM and cNIRS (Group 3). A survey called NASA Task Load Index will be used to study HCPs workload. On a small number of teams, the investigators will also track where the leader of the team is looking using eye-tracking glasses, how stressed the leader is by measuring their heart rate, skin sweat, and pupil dilation. Finally, the investigators will collect some information about the baby's resuscitation and hospital stay.

DETAILED DESCRIPTION:
The investigators aim to study 93 resuscitations of very preterm infants (23+0-31+6 weeks), in consecutive groups of 31. First, as a baseline, 31 infants will be resuscitated using the standard approach, with vital signs monitoring only. Subsequently, 31 infants will be resuscitation with the addition of Respiratory Function Monitor (RFM) to measure VT. Finally, 31 infants will be resuscitated using vital signs monitor, RFM, and cerebral near-infrared spectroscopy (NIRS). Study participants will be health care providers, and the primary endpoint is based on the recruitment of 93 team leaders (31 in each group). Other team members will also be recruited, to an estimate of 3-5 team members per resuscitation in total (N=279 to 465). Throughout the study, HCPs will be trained to incorporate the use of RFM and NIRS in their resuscitation decision-making, using a combination of weekly in-situ simulations and incorporation of NIRS and RFM teaching into ongoing resuscitation team educational sessions and practice updates. Suggested tidal volume and NIRS goals will be posted as cognitive aids in the resuscitation rooms throughout the study. This sequential approach will allow for resuscitation teams to become acclimatized to the use of RFM and NIRS as routine practice. The sequential approach will also allow the investigators to study time-based changes in perceived mental workload as teams acclimatize to the use of additional monitoring.

After each resuscitation, all team members involved will be asked to complete a brief workload questionnaire (NASA-Task Load Index), which will be linked to the resuscitation. Resuscitations will be video-recorded for analysis of i) resuscitation steps required (e.g. basic steps, bag-mask ventilation, endotracheal intubation, chest compressions, medications), and ii) frequency of use of additional monitoring data (RFM, NIRS) for decision-making. In a subset of resuscitations, the team leader will also be equipped with eye-tracking glasses to record visual attention and pupillary dilatation, and Empatica wristband to record the team leader's heart rate and EDA. Parents of the infants will then be approached for permission to collect more detailed information for the infant's resuscitation and subsequent hospitalization.

Data will be analyzed to compare i) team leader subjective mental workload, ii) composite team mental workload, iii) other workload measures (physical demand, temporal demand, performance, effort, frustration), iii) percentage of visual attention focused on infant, monitoring devices, and other HCPs, iv) frequency of visual access to each monitor display type (vital signs, RFM, NIRS), iv) respiratory function (VT, PIP), v) cerebral NIRS, vi) time to placement of monitoring probes (ECG leads, pulse oximetry, cerebral NIRS), vii) time to first reading for each monitoring device, and viii) time to target HR and SpO2. The primary outcome will be the perceived mental workload of the team leader. Data will be compared between the three groups. In addition, time-dependent changes in team leader and composite mental workload will also be analyzed using a run chart approach. Deferred consent will be obtained from each infant's parents / guardians for collection of hospital course data including: i) incidence of intraventricular hemorrhage, ii) respiratory supports needed, iii) bronchopulmonary dysplasia at 36 weeks, iv) death / survival to discharge.

ELIGIBILITY:
Inclusion Criteria:

* HCPs participating in resuscitations of very preterm infants (23+0-31+6 weeks) at the Royal Alexandra Hospital Neonatal Intensive Care Unit (NICU), a Level III NICU will be included.
* Multiple gestations will be analyzed individually as separate resuscitations. HCPs will include different levels of experience and different disciplines (registered nurses, advance practice nurses, respiratory therapists, neonatal nurse practitioners, pediatric residents, neonatal fellows, clinical associates, and neonatal consultants).
* All HCPs who participate in the resuscitation, regardless of role, will be eligible for completion of NASA-TLX surveys.
* Participants who act as team leader will be eligible to be fitted with eye-tracking glasses to record their visual attention and Empatica E4 wristbands to measure physiological stress measurements.
* For resuscitated infants, hospital outcomes will be included with parental consent.

Exclusion Criteria:

* Teams involved in the resuscitation of infants born with congenital malformations, or involved in the care of infants for whom active resuscitation is not planned (i.e., comfort care only for periviable gestations) will be excluded.
* Teams who do not consent to participate will also be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Team Leader's NASA Task Load Index (NASA-TLX) Mental Demand | Immediately post resuscitation
  Team leader's subjective mental demand as reported by the NASA Task Load Index

SECONDARY OUTCOMES:
Composite team mental workload | Immediately post resuscitation
  Team members combined mental workload as measured by NASA Task Load Index
Team Leader Visual Attention Distribution | During resuscitation
  Percentage of visual attention focused on infant, monitoring devices, and other health care provider as measured by mobile eye-tracking
Frequency of visual fixation to monitoring equipment Visual Access to each monitor display type (vital signs, RFM, NIRS) | During resuscitation
  Frequency of visual fixation to vital signs monitor, Respiratory function monitoring (RFM) screen, and Near Infrared Spectroscopy (NIRS) screen as measured by eye-tracking
Time to achieving target heart rate (HR) and oxygen saturation (SpO2) | During resuscitation
  Time to achieving target HR and SpO2 for age during resuscitation
Survival to 36 weeks | 36 weeks
  Survival to 36 weeks
Severe Intraventricular hemorrhage | 36 weeks
  Grade III or Grade IV Intraventricular hemorrhage
Severe Bronchopulmonary Dysplasia | 36 weeks
  Need for ≥30% oxygen and/or positive pressure, (PPV or NCPAP) at 36 weeks PMA or discharge, whichever comes first.
Team Leader's heart rate during resuscitation | During resuscitation
  Team Leader's median heart rate during resuscitation as an indicator of stress
Team Leader's electrodermal activity | During resuscitation
  Team Leader's electrodermal activity as an indicator of stress
Time to apply all probes | During resuscitation
  Time to apply the probes as needed by the group (SpO2, ECG, NIRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided